CLINICAL TRIAL: NCT02973308
Title: The Inter and Intra Reliability of Cardiopulmonary Exercise Testing in Abdominal Aortic Aneurysm Patients
Acronym: CPEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 199037
Record Dates: First submitted 2016-10-19; First posted 2016-11-25 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Observer Variation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treadmill-Test operator A (Other): Randomised to motorised treadmill group A for inter reliability, observer A will perform both exercise tests
  Interventions: Other: Observer
- Treadmill-Test operator B (Other): Randomised to motorised treadmill group B for intra reliability, observer A will perform one exercise test, followed by observed B
  Interventions: Other: Observer
- Cycle-Test operator A (Other): Randomised to cycle group B for inter reliability, observer A will perform both exercise tests
  Interventions: Other: Observer
- Cycle-Test operator B (Other): Randomised to cycle group B for intra reliability, observer A will perform one exercise test, followed by observed B
  Interventions: Other: Observer

INTERVENTIONS:
Other: Observer — Observer A and observer B

SUMMARY:
Exercise testing is commonly being used in patients before surgery to test their overall fitness. One group it is being used in is patients who have an enlarged blood vessel in their stomach. This is known as an abdominal aortic aneurysm. The exercise test used is known as a cardiopulmonary exercise test as it looks at both heart and lung function at the same time. Whilst this test is commonly used there have been no studies (to date) which have looked at how reliable this test is; this means how well the investigators can obtain the same (or very similar) results after multiple tests. The investigators would like to test this reliability both between patients and the clinicians performing the testing.

DETAILED DESCRIPTION:
Background Research:

The definition of an 'aneurysm' is permanent, localised dilatation of a blood vessel or heart chamber. The abdominal aorta is the largest blood vessel in the human body and usually has a diameter of 1.8 -2.0 centimetres (cm), dependant on age, sex and body habitus. Aortic dilatation is generally classed as an 'aneurysm' when dilation of the vessel is 1.5 times the normal size. An abdominal aortic aneurysm (AAA) affects any part of the aorta below the diaphragm with 80 % typically being found between the renal artery and aortic bifurcation.

Risk Factors There are many factors that relate to the development of AAA. Gender is one of the biggest non-modifiable risk factors, as an AAA is four to six times more likely in males compared with females. Furthermore, the development of AAA in females occurs approximately ten years later than males. The risk of AAA also increases if there is family history of the disease, especially if the relative is first degree. There is also evidence to suggest there is an association between AAA and coronary heart disease. Hypertension has also been found to closely correlate with the development of AAA. Additionally, there is also a strong link between smoking and the likelihood of AAA development. Conversely, whilst the risk of AAA development in women is less than men, women have been shown to be more vulnerable to developing AAA than their male counterparts. The risk of AAA's also increases after the age of 65 years.

If AAA are left undetected or untreated there is an increase in the likelihood of a rupture occurring. This causes critical internal bleeding and often results in death. Rupture of AAA is the cause of approximately 6000 deaths per year in the United Kingdom. Figures between 1997- 2005 have shown a decrease in mortality but this is due to an earlier detection (of around five to ten years). The likelihood of rupture increases due to age, sex, smoking, hypertension and size and growth rate of the aneurysm. The size of the aneurysm is the strongest predictor of risk of rupture, smoking also contributes to an acceleration in expansion rate.

Ultrasound Screening:

Ultrasound screening is the preferred tool in identifying and monitoring the development of AAA as it is highly sensitive, cost effective and a non-invasive tool. The National Institute of Clinical Excellence (NICE) guidelines recommend that the National Health Service (NHS) offers ultra-sonographic screening to all males age 65 or over. The ultrasound scan enables the medical screener to determine the size of the abdominal aorta. According to the NICE (1.3) guidelines AAA are categorised by size, with a diameter of less than three cm being classified as normal with no follow up required. Patients who have an aneurysm diameter of between 3- 4.4 cm are re-scanned yearly, with those between 4.5 -5.4 cm being rescanned quarterly (every three months). AAA patients who have a diameter greater than 5.4 cm are referred to a vascular consultant for diagnosis and treatment. An AAA can be either true or false, with true aneurysms more commonly found. True aneurysms; involve three layers of the blood vessel walls Intima, Media and Adventitia, whereas false aneurysms are essentially a haematoma that forms outside the vessel wall.

Surgical management of AAA:

Following the diagnosis of a large AAA there are two possible medical surgical interventions, open or endovascular repair (EVAR).Open repair is considered to be a major surgical procedure and because of the possible complications preoperative assessment has to be carefully managed. There are three approaches whilst performing AAA laparotomy, transverse incision, longitude midline incision and retroperitoneal approach. The aortic segment is replaced by a prosthetic graft. After the operation patients are often monitored in intensive care unit (ICU) on average remain in hospital between seven to fourteen days. EVAR on the other hand is less invasive procedure, less painful and has a shorter stay in hospital and often does not require stay in ICU. EVAR gains access though the femoral artery and inserts a sent graft inside the abdominal aneurysm.

Preoperative Risk Management:

Surgeons base the decisions for operating on two major factors, firstly the risk of rupture, and secondly the diameter of the aneurysm and the growth rate. Before surgery the vascular consultant will subject the patient to a preoperative functional capacity assessment (FCA). The surgeons use FCA to establish if there are any potential operative and postoperative risks. Patients often have other comorbidities so the risk of operating may outweigh the potential benefits, therefore increasing the risk of premature mortality. The use of FCA has become an important screening tool in evaluating the fitness of AAA patients, serving as a good indictor to the risk of surgery and postoperative recovery. There are various ways to test FCA (step test, spirometry and cardiopulmonary exercise testing etc.) however, more recently cardiopulmonary exercise testing has been described as preferable tool in evaluating AAA patient's functional capacity.

Cardio pulmonary exercise testing:

It is widely accepted that a cardio-pulmonary exercise test (CPEX) is the 'gold standard' of FCA. Furthermore, CPEX is a non-invasive, cost effective and objective. It has been used for many years in elite sporting performance for research and screening and is now becoming increasingly utilised in clinical environments. CPEX testing allows clinicians to perform a controlled exercise test in a safe environment. It involves the measurement of a number of physiological parameters, as well as respiratory and cardiac monitoring.The basic underlying physiological principles underlying a CPEX is that it measures the efficiency and capacity of the oxygen-transport system; it also examines an individual's ability to exercise and the cardiovascular responses to variable levels of exertion. A CPEX provides breath by breath analysis and provides several important outcomes. These are; (1) VO2 MAX, (2) VeO2, (3) VECO2, (4)anaerobic threshold (AT), (5) respiratory exchange ratio, (6) time to AT and (7) total time tolerated are the variables that are obtained.

Anaerobic threshold (AT):

At the beginning of exercise, adenosine trisphosphate-creatine phosphate provides immediate energy required by the working muscles. As exercise continues cardiac output increases providing the working muscles with increased blood flow. As exercise levels rise, the workload of the muscles also rises requiring more blood flow and oxygen to be delivered. The oxygen demand is met by an increase cardiac output and lung ventilation. As the exercise continuous to become more strenuous, the muscle demand will begin to exceed the rate of oxygen delivery by the respiratory system. At this point the main fuel glucose is metabolised into lactic acid. This dissociates to lactate and hydrogen ions (H+) resulting in acidosis, which is the marker known as the Anaerobic Threshold (AT). The most common way of measuring the AT non-invasively is the V-slope method see figure 1.

This can be explained via the following:

As a participant begins incremental exercise their expired minute volume (VE) increases linearly with their oxygen consumption (VO2) and carbon dioxide consumption (VCO2). H+ are produced via anaerobic metabolism which is buffered by bicarbonate (HCO3-) and produces carbon dioxide (CO2). This is washed out in the lungs and is measured via the breath by breath analysis in the expired air. As VCO2 rises disproportionately to VO2, it allows the clinician to determine the AT; this is achieved by plotting VCO2 against VO2. Linear regression lines are drawn through the upper and lower curve and the point of intersection indicates where VCO2 increased disproportionately to VO2 and hence is estimated to be the AT.

An individual's aerobic capacity is known as their VO2MAX. The most common way of measuring a person VO2 max is an incremental exercise test either performed on a motorized treadmill or cycle-ergometer, measured in millilitres per kilogram per minute (ml.kg.min). The aerobic capacity can be affected by factors such as gender, genetics, body composition and age. A healthy 20-25 year old male has an average VO2 max of 42.5 - 46.4 ml.kg.min, whereas a healthy female of the same age has an average of 33 - 36.9 ml.kg.min. There is approximately ten percent drop with aerobic capacity every decade (dependent on fitness). For patients with AAA it is suggested that they should achieve and a threshold (AT) value above 10.2 ml.kg.min for open repair or above 8.2 for EVAR. They should also achieve a VO2MAX value above 15 ml.kg.min. Values lower than this can increase the risk of postoperative mortality (within 30 days).

Whilst there have been numerous studies into the importance of a CPEX, there have been no studies to date which have determined the Inter and Intra reliability of this test in the AAA population.

Aim:

The aim of this study is therefore to determine the Inter and Intra reliability of CPEX testing on both a cycle- ergometer and motorised treadmill in patients with abdominal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* • Must be over the age of 45

  * The patients must have the ability to walk unaided
  * Must be considered for open or endovascular repair
  * Have an AAA diameter of 5.4 cm or over.
  * English speaking and able to follow simple protocol instructions

Exclusion Criteria:

* • Active cancer treatment.

  * Patients whom are not able to give informed consent
  * Severe cardiovascular, musculo-skeletal or pulmonary illness precluding ability to partake in CPEX testing.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07-03 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Anaerobic threshold | Up to One week
  The anaerobic threshold is a physiological measurement which is generated via breath by breath analysis and determined by the v-slope method as described in the summary.

SECONDARY OUTCOMES:
Minute ventilation | Up to One week
  Physiological measurement, computer generated via the breath by breath analysis
Respiratory exchange ratio | Up to One week
  Physiological measurement, computer generated via the breath by breath analysis
Total time of exercise | Up to One week
Quality of life Questionnaire | Up to One week
Time to anaerobic threshold | Up to One week
Maximal oxygen uptake | Up to One week
  Physiological measurement, computer generated via the breath by breath analysis

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Harwood, MSc, Principal Investigator — AVSU Hull Royal Infirmary
Locations (1):
- Academic Vascular Surgery Unit, Vascular Laboratory, Alderson House, Hull Royal Infirmary, Hull, East Riding Of Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share participant data

REFERENCES:
- [Result] Harwood AE, Pymer S, Hitchman L, Totty J, Wallace T, Smith GE, Carradice D, Carroll S, Chetter IC. The Intrarater and Interrater Reliability of Measures Derived from Cardiopulmonary Exercise Testing in Patients with Abdominal Aortic Aneurysms. Ann Vasc Surg. 2019 Apr;56:175-182. doi: 10.1016/j.avsg.2018.08.087. Epub 2018 Nov 23. PMID 30476603